CLINICAL TRIAL: NCT06920615
Title: Stereotypi in Motor-, Vocal- and Feeding Behaviors: Novel Extensions to Adults
Brief Title: Stereotypic Behaviors and Feeding Difficulties in Adults With Developmental Disabilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Petur Ingi Petursson, Principal investigator, Oslo University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 830334; 25/05900 (Other: Oslo University Hospital)
Record Dates: First submitted 2025-04-08; First posted 2025-04-10 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Harmful Stereotypies; Feeding Difficulties
Keywords: Feeding difficulties, stereotypic behavior, challenging behavior, autism, developmental disabilities
MeSH Terms: conditions — Stereotypic Movement Disorder; Autistic Disorder; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: The research utilizes single-case experimental designs for each individual participant
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intake refusal (Experimental): Intervention
  Interventions: Behavioral: Fading and chaining combined with differential reinforcement
- Slow pace of self-feeding (Experimental): Intervention
  Interventions: Behavioral: Differential reinforcement of high rate
- Debilitating stereotypi (Experimental): Intervention
  Interventions: Behavioral: Response interruption with redirection; Behavioral: Chained schedules

INTERVENTIONS:
Behavioral: Fading and chaining combined with differential reinforcement — Intervention Treatment will involve backward chaining, fading and differential reinforcement.
  Arms: Intake refusal
Behavioral: Differential reinforcement of high rate — This will be identical to baseline, except a DRH will be introduced: The participant will be instructed to complete his whole meal within set time criteria to receive an identified reinforcer.
  Arms: Slow pace of self-feeding
Behavioral: Response interruption with redirection — RIRD involves physically blocking a movement from occurring using the least amount of physical contact for max 3 s, and then redirecting behavior to an ongoing activity or movement. Stereotypi that is verbal or not possible to block physically will involve a demand to answer a verbal question or a motor task that sufficiently interrupts the behavior and then redirecting.
  Arms: Debilitating stereotypi
Behavioral: Chained schedules — The following procedures are based on Slaton et al. (2016): At the start of each session, the candidate or therapist will hold up the red card, prompt the participant to touch the card, while saying "we are in red now, time to work". The participant will have to perform age- or function appropriate tasks without stereotypi to gain access to the green phase. Demand will be designated with a token economy, where each token represents completion of a certain amount of task-related responses. The participant will not be prompted to perform the tasks. If the participant makes an error in a task (e.g. answer a math question incorrectly), this will lead to an error correction and no token will be presented. If stereotypi occurs, it will be blocked for up to 3 s, and then all demands will be reset by removing all earned tokens.
  Other Names: Differential reinforcement utilizing access to stereotypi
  Arms: Debilitating stereotypi

SUMMARY:
Adults with developmental disabilities (DD) and autism represent a vulnerable demographic that transitions into adulthood with diverse etiologies, exhibiting a significantly higher prevalence of various challenging behaviors. These problematic behaviors can lead to adverse health outcomes and a diminished quality of life. Addressing these issues often necessitates an interdisciplinary approach to continuity of care, focusing on enhancing functional skills, empowerment, and independence, as well as preventing and mitigating challenging behaviors. The current research proposal comprises of three studies designed to evaluate the efficacy of behavioral interventions for problematic behaviors in adults with DD and autism. If left unaddressed, these behaviors may worsen over time, potentially hindering community involvement, educational opportunities, and employment prospects. These include harmful stereotypies and feeding difficulties.

DETAILED DESCRIPTION:
Study 1: A behavioral intervention of food refusal in adults with developmental disabilities

Feeding disorders are common in both children and adults with DD. Among the most serious of these is the total refusal to consume food and liquid, which may present a life-threatening or severely debilitating condition. The evidence base for interventions for adults with DD and food refusal is severely limited or lacking to my knowledge. One notable exception is a study by Kitfield and Masalsky (2000), who treated a woman aged 22 using a behavioral intervention consisting of negative reinforcement in the form of escape from food as well as to other areas, which resulted in impressive weight gains during treatment and follow-up. The lack of empirically supported treatment for food refusal in adults with DD may be because food-related issues usually have an early onset and are, therefore, more often diagnosed and treated in children. Additionally, some treatments may be viewed as more invasive when applied to adults. For example, escape extinction is the most empirically supported treatment component for food refusal and selective eating among children with DD. However, implementing escape extinction in an adult may be ethically questionable because of its invasive nature, which is practically challenging or dangerous, especially when other problem behaviors are present.

In a study by Hagopian et al. (1996), total food and liquid refusal in a 12-year old boy with autism was treated with backward chaining, fading, and activity reinforcement, which successfully resulted in drinking from a cup generalized to his living unit. Fading and differential reinforcement may have an ethical and intuitive appeal when treating food and liquid refusal in adults with DD and may therefore be accepted by caregivers and adults with DD. This is because it involves gradual re-introduction of oral intake and the use of positive reinforcement. In addition, research has demonstrated that stimulus fading may render escape extinction unnecessary. Therefore, there is a need to extend the use of such procedures to adults with food and/or liquid refusal.

Study 2: A behavioral intervention of slow eating in adults with DD

Individuals with DD often require considerably more time to complete tasks of daily living than their neurotypical peers do. When slow responding becomes excessive, it may be a barrier in daily living as self-care, and finishing meals in time before scheduled events may lead to missed activities or services, family stress, and logistical challenges. Such slowness has been hypothesized to result from neurological impairments causing a slow motor response, a secondary symptom of obsessive compulsive disorder, or as a primary feature, an operant modifiable by its consequences.

Slow responding has been the subject of three empirical investigations in the behavioral literature, with two children and one adult. In all cases, the researchers utilized positive reinforcement to accelerate slow responses. Fjellstedt and Sulzer-Azároff (1973) used a differential reinforcement of low response latencies (DRL) for the following five different types of instructions to perform tasks, resulting in a substantial improvement in the speed of response. Tiger et al. (2007) increased the slow response of an adult male with Asperger's syndrome with a DRL, which resulted in a clinically significant increase in the response to two tasks. Girolami et al. (2008) utilized differential reinforcement of high rate (DRH) to increase the rate of independent bites by a child participant with ADHD and several medical issues. This procedure results in an increased rate of self-feeding. We plan to systematically replicate a DRH procedure for adults suffering from slow-feeding difficulties, with modifications involving the use of changing criteria for reinforcement.

Study 3: A behavioral treatment of debilitating stereotypy in adults, comparing response interruption with redirection and chained schedules

Stereotypy refers to behavior topographies in individuals with autism and DD that are invariable, repeating, meaningless, or out of context. These topographies can present a considerable amount of distress for the individuals and their family members as it may be a barrier for habilitation, independent living and learning. Because the majority of researched stereotypi in individuals with autism have automatic reinforcement as its function, a new strategy for functional analysis (FA) of stereotypi involves pre-treatment screening for automatic reinforcement.

Function-based treatment of automatically maintained stereotypy is particularly challenging because reinforcers are not easily manipulated or extinguished. Physically preventing stereotypi in adults may be practically challenging, especially because it may elicit emotional or aggressive behavior. For example, response blocking has been documented to reduce automatically maintained pica but increase aggressive behavior. Research has shown that when stereotypi are both blocked and redirected toward an ongoing behavior, aggressive behavior does not increase. A treatment procedure for automatically maintained stereotypi, called response interruption with redirection (RIRD), involves interrupting each instance of stereotypi and redirecting behavior to an ongoing task or appropriate behavior. RIRD has received extensive empirical support from child participants for reducing stereotypi, but has not been researched in adults. Another treatment procedure that has recently received increased attention in behavioral literature is chained schedules (CS), often contrasted with multiple schedules (MS), both of which are different procedures for programming stimulus control over stereotypi. MS involves the use of discriminative stimuli (SD/S+ vs. SΔ/S-) for different treatment components, where in one phase, all instances of stereotypi are blocked in the presence of S- (e.g., at red card), while in the presence of S+ (e.g., a green card), all instances of stereotypi are allowed. However, no reinforcement contingency was programmed. On the other hand, CS also involves blocking stereotypi in the presence of S-, but providing contingent access to stereotypi from one component (red card/ S-) to the other (green card/ S+) contingent upon the absence of stereotypi. Therefore, alternation between the two components depends on the performance of one of the components. When compared to MS, most empirical demonstrations favor CS, both in terms of the reduction of stereotypi and an increase in adequate item engagement. As pointed out by Sloman et al. (2022), autism advocates view access to "stimming" as a means for individuals with autism to self-sooth and regulate emotions, and may therefore be more preferred. However, the CS procedure is more complicated than the RIRD procedure (see below). In addition, the RIRD does not program a differential reinforcement of alternative responses. CS may, therefore, be preferred by adults and caregivers in that it targets increasing adaptive responses. However, some treatment settings may favor RIRD over CS because of its ease of implementation. An interesting question is whether caregivers and clients provide different answers to these questions. Therefore, the current research question concerns a) the efficacy of RIRD as compared to CS, both in terms of behavior reduction and treatment duration, b) client vs. caretaker preference for either treatment procedure, c) extension of these two empirically supported treatments to adult participants, and d) generalization to the most problematic settings in daily life.

[PP2]Hope this clears it up

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited through referrals at the Department of Neurohabilitation, or from other hospitals in the Oslo Region.
* be 18 years or older,
* have a DD, autism spectrum disorder or a PDD-NOS diagnosis
* and be referred to the specialist habilitation service for adults.

Exclusion Criteria:

* If there are medical causes of the participant's behavioral problem or
* a reasonable possibility that the referred problem is caused by medical variables
* if the client participant receives communal care services and if those are not in accordance with Norwegian standards of services for individuals with DD.
* This could include inappropriate staff-to-client ratio,
* lack of stimulating activities,
* or if on-site training is insufficient.
* the exclusion criteria do not exclude health care from The Oslo University Hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-04-08 (Estimated); Primary Completion 2030-08-26 (Estimated); Study Completion 2030-08-26 (Estimated)

PRIMARY OUTCOMES:
Frequency recording | Each experimental phase will last until there is a stable-state performance of the target behavior, typically within 4-8 weeks.
  Each target behavior in the study will be measured with a frequency recording and graphed as behavior change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Petur I Petursson, MS, BCBA, Principal Investigator — Oslo University Hospital; Sigmund Eldevik, PhD, BCBA-D, Study Chair — Oslo Metropolitan University
Locations (1):
- Department of Neurohabilitation, Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams, E.W., Seiverling, L.J., & Field, D.G. (2014). Feeding problems. In: P. Sturmey & R. Didden (Eds.), Evidence-Based Practice and Intellectual Disabilities (pp. 198-213). Wiley Blackwell.
- [Background] Volkert, V.M., Patel, M.R., Peterson, K.M. (2016). Food refusal and selective eating. In: Luiselli, J. (ed) Behavioral Health Promotion and Intervention in Intellectual and Developmental Disabilities. Evidence-Based Practices in Behavioral Health. Springer, Cham. https://doi.org/10.1007/978-3-319-27297-9_7
- [Background] Ratnasuriya RH, Marks IM, Forshaw DM, Hymas NF. Obsessive slowness revisited. Br J Psychiatry. 1991 Aug;159:273-4. doi: 10.1192/bjp.159.2.273. PMID 1773246
- [Background] Kitfield EB, Masalsky CJ. Negative reinforcement-based treatment to increase food intake. Behav Modif. 2000 Sep;24(4):600-8. doi: 10.1177/0145445500244007. PMID 10992614
- [Background] Association of Professional Behavior Analysts. (2009). The use of restraint and seclusion as interventions for dangerous and destructive behaviors. www.apbahome.net/Restraint_Seclusion%20.pdf
- [Background] Kazdin (2021). Single-case research designs: Methods for clinical and applied settings. Oxford University Press.
- [Background] Jarness, M., Petursson, P.I. & Eldevik, S. (2019). Trening av verbale operanter og differensiell forsterkning fører til økning i passende vokalisering og reduksjon i upassende vokalisering: Et kasus studie basert på en funksjonell analyse. Norsk Tidsskrift for Atferdsanalyse, 46, 71-83.
- [Background] Iwata BA, Dorsey MF, Slifer KJ, Bauman KE, Richman GS. Toward a functional analysis of self-injury. J Appl Behav Anal. 1994 Summer;27(2):197-209. doi: 10.1901/jaba.1994.27-197. PMID 8063622
- [Background] Hagopian LP, Kurtz PF, Bowman LG, O'Connor JT, Cataldo MF. A Neurobehavioral Continuum of Care for Individuals with Intellectual and Developmental Disabilities with Severe Problem Behavior. Child Health Care. 2023;52(1):45-69. doi: 10.1080/02739615.2021.1987237. Epub 2022 Jan 25. PMID 36643575
- [Background] Hagopian LP, Farrell DA, Amari A. Treating total liquid refusal with backward chaining and fading. J Appl Behav Anal. 1996 Winter;29(4):573-5. doi: 10.1901/jaba.1996.29-573. PMID 8995838
- [Background] Grinblat N, Rosenblum S. Why are they late? Timing abilities and executive control among students with learning disabilities. Res Dev Disabil. 2016 Dec;59:105-114. doi: 10.1016/j.ridd.2016.07.012. Epub 2016 Aug 12. PMID 27525557
- [Background] Fjellstedt N, Sulzer-Azaroff B. Reducing latency of a child's responding to instructions by means of a token system. J Appl Behav Anal. 1973 Spring;6(1):125-30. doi: 10.1901/jaba.1973.6-125. PMID 16795384
- [Background] Fisher W, Piazza CC, Bowman LG, Hagopian LP, Owens JC, Slevin I. A comparison of two approaches for identifying reinforcers for persons with severe and profound disabilities. J Appl Behav Anal. 1992 Summer;25(2):491-8. doi: 10.1901/jaba.1992.25-491. PMID 1634435
- [Background] Borrero, C. S., Schlereth, G. J., Rubio, E. K., & Taylor, T. (2013). A comparison of two physical guidance procedures in the treatment of pediatric food refusal. Behavioral Interventions, 28, 261-280. https://doi.org/10.1002/bin.1373